CLINICAL TRIAL: NCT04992780
Title: A Randomized Phase II Trial of Hypo-fractionated Intensity-Modulated Radiation Therapy (IMRT) Utilizing 2.5 Gy/Fraction Versus (VS) Standard-Fractionated IMRT, Concurrent With Carboplatin/Paclitaxel and Followed by Consolidation Durvalumab, for Subjects With Stage 2A/B Non-Small Cell Lung Cancer
Brief Title: Comparing Hypo-fractionated Intensity- Modulated Radiation Therapy to Standard- Fractionated IMRT Along With Chemotherapy and Immunotherapy for Non-Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT-2021-LU-HypoIMRT
Record Dates: First submitted 2021-07-28; First posted 2021-08-05 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Non Small Cell Lung Cancer Stage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Hypo-Fractionation (Experimental): Participants will receive one fraction of radiation therapy a day for 5 days each week for 5 weeks along with weekly chemotherapy with Paclitaxel 45 milligram per meter squared (mg/m2) through intravenous (IV)infusion for 1 hour followed by Carboplatin area under the curve (AUC) 2 IV for 30 minutes for approximately 5 or 6 weeks. Once complete, participant will receive Durvalumab, 1500 mg, IV every 4 weeks for 12 months.
  Interventions: Radiation: Hypo-Fractionation
- Standard-Fractionation (Active Comparator): Participants will receive one fraction of radiation therapy a day for 5 days each week for 6 weeks along with weekly chemotherapy with Paclitaxel 45 milligram per meter squared (mg/m2) through intravenous (IV)infusion for 1 hour followed by Carboplatin AUC 2 IV for 30 minutes for approximately 5 or 6 weeks. Once complete, participant will receive Durvalumab, 1500 mg, IV every 4 weeks for 12 months.
  Interventions: Radiation: Standard-Fractionation

INTERVENTIONS:
Radiation: Hypo-Fractionation — 62.5 Gy in 25 fractions of 2.5 Gy/fraction
  Arms: Hypo-Fractionation
Radiation: Standard-Fractionation — 60 Gy in 30 fractions of 2 Gy/fraction
  Arms: Standard-Fractionation

SUMMARY:
The hypothesis for this study is that hypofractionated IMRT to 62.5 Gy in 25 fractions (2.5 Gy/fraction) with concurrent carboplatin and paclitaxel, followed by maintenance durvalumab will improve locoregional control at 18 months by 10% compared to standard-fractionated chemo-IMRT/durvalumab. A modest improvement in locoregional control (LRC) was selected as a target which could merit further study of this hypofractionated IMRT regimen in a Phase III trial

ELIGIBILITY:
Inclusion Criteria:

* Ability of participant OR Legally Authorized Representative (LAR) to understand this study, and participant or LAR willingness to sign a written informed consent
* Males and females age ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0 - 2
* Measurable disease by RECIST 1.1
* Women of childbearing potential must have a negative serum pregnancy test within one month prior to initiating treatment
* Pathologically proven diagnosis of Stage IIIA or IIIB non-small cell lung cancer (NSCLC)
* No Positron Emission Tomography (PET)/CT evidence of metastatic disease
* An MRI of the brain with contrast excluding intracranial metastatic disease (or CT with contrast if MRI is medically contraindicated). An MRI without contrast is only permitted if the subject cannot have contrast for medical reasons
* If a pleural effusion is present, it must be tapped and confirmed to be cytologically negative. If an effusion is deemed too small to safely tap, the subject will be eligible
* Women of child-bearing potential and men with partners of child-bearing potential must agree to practice sexual abstinence or to use the forms of contraception listed in Child-Bearing Potential/Pregnancy section for the duration of study participation and for 90 days following completion of therapy
* Adequate organ function per laboratory results

Exclusion Criteria:

* Current or anticipating use of other anti-neoplastic or investigational agents while participating in this study
* Diagnosed with a psychiatric illness or is in a social situation that would limit compliance with study requirements
* Evidence of severe or systemic disease (e.g., unstable or uncompensated respiratory, cardiac, hepatic, or renal disease) that would interfere with study protocol as judged by the investigator
* Is pregnant or breastfeeding
* Active connective tissue disorders, such as active lupus or scleroderma
* Known Acquired Immune Deficiency (HIV (+)/AIDS)
* Has a known allergic reaction to any excipient contained in the study drug formulations
* Active Grade 3 (per the NCI CTCAE, Version 5.0) or higher viral, bacterial, or fungal infection within 2 weeks prior to the first dose of study treatment
* Prior thoracic radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-02-25 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Locoregional control (LRC) | From enrollment for up to 7.5 years
  RECIST 1.1

SECONDARY OUTCOMES:
Acute toxicities | From enrollment for up to 7.5 years
  CTCAE v. 5.0
Late toxicities | From enrollment for up to 7.5 years
  CTCAE v. 5.0
Progression free survival (PFS) | From enrollment for up to 7.5 years
  RECIST 1.1
Overall survival (OS) | From enrollment for up to 7.5 years
  Kaplan-Meier
Measuring the Impact of Treatment on the Quality of life (QOL) | From enrollment for up to 7.5 years
  EORTC Quality of Life Questionnaire (QLQ)-C30
Measuring the Impact of Treatment on the Quality of life (QOL) | From enrollment for up to 7.5 years
  QLQ-Lung Cancer (LC)29

CONTACTS AND LOCATIONS:
Overall Officials: Krishna Reddy, MD, PhD, Principal Investigator — University of Kansas Medical Center
Locations (6):
- United States (6):
  - The University of Kansas Cancer Center, Westwood Campus, Kansas City, Kansas
  - The University of Kansas Cancer Center, Overland Park Clinic, Overland Park, Kansas
  - KUCC MCA- TUKHS, Saint Francis Hospital, Topeka, Kansas
  - The University of Kansas Cancer Center, North Clinic, Kansas City, Missouri
  - The University of Kansas Cancer Center, Lee's Summit Clinic, Lee's Summit, Missouri
  - University of Kansas Cancer Center, North Kansas City Hospital, North Kansas City, Missouri

IPD SHARING:
Plan to Share IPD: Undecided